CLINICAL TRIAL: NCT02126813
Title: Urinary Bladder Catheterization in Fast-track Hip and Knee Arthroplasty - What is the Optimal Bladder Volume? A Randomized, Controlled Study
Brief Title: When to Perform Bladder Catheterization in Fast-track Hip and Knee Arthroplasty
Acronym: POUR-RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Lundbeck Foundation (Other)
Responsible Party: Principal Investigator, Lars Bjerregaard, M.D., Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: POUR-RCT
Record Dates: First submitted 2014-04-24; First posted 2014-04-30 (Estimated); Last update posted 2015-10-28 (Estimated); Status verified 2015-10

CONDITIONS: Postoperative Urinary Retention (POUR)
Keywords: Postoperative urinary retention; Fast-track total hip (THA) and knee arthroplasty (TKA); Urinary bladder volume

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 500 ml. (Active Comparator): A bladder volume of 500 ml. or more, and incapability of voluntary micturition, is used as interventional threshold for urinary bladder catheterization.
  Interventions: Procedure: Current used interventional threshold for urinary bladder catheterization (500 ml); Device: Intermittent bladder catheter
- 800 ml (Experimental): A bladder volume of 800 ml. or more, and incapability of voluntary micturition, is used as interventional threshold for urinary bladder catheterization.
  Interventions: Procedure: increased interventional threshold for urinary bladder catheterization (800 ml); Device: Intermittent bladder catheter

INTERVENTIONS:
Procedure: increased interventional threshold for urinary bladder catheterization (800 ml)
  Arms: 800 ml
Procedure: Current used interventional threshold for urinary bladder catheterization (500 ml)
  Arms: 500 ml.
Device: Intermittent bladder catheter

SUMMARY:
Approximately 40 % of all patients undergoing fast-track total hip or knee arthroplasty needs intermittent bladder catheterization after surgery, as they are transient incapable of voluntary bladder emptying (postoperative urinary retention - POUR). The currently used interventional threshold for urinary bladder catheterization are a bladder volume of approximately 500 ml., but no evidence exists for this threshold. At the same time, the current knowledge suggest, that a bladder volume up to 1000 ml. for 2-4 hours are safe in humans, and as the use of urinary bladder catheterization are increasing the risk of complications, the investigators are hypothesizing that increasing the interventional threshold for urinary bladder catheterization after fast-track total hip or knee arthroplasty, will reduce the number of patients needing urinary bladder catheterization, without increasing the incidence of urological complications - including urinary tract infections.

ELIGIBILITY:
Inclusion Criteria:

* planned for elective total hip or knee arthroplasty
* given written informed consent for participation

Exclusion Criteria:

* can't co-operate to participation
* can't speak or understand danish
* preoperative use of urinary bladder catheterization
* using haemodialysis
* previous cystectomy
* need for permanent urinary bladder catheter during surgery (decided by anaesthesiologist and/or surgeon)
* Pregnant or given birth within the last 6 months

Ages: 18 Years to 125 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Actual)
Dates: Start 2014-05; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Number of patients receiving postoperative urinary bladder catheterization | Patients will be followed from end of surgery to their first voluntary micturition, expectably within a mean period of twelve hours

SECONDARY OUTCOMES:
Incidence of urinary tract infections | within the first 30 days after surgery
Number of voiding difficulties acquired postoperatively | within the first 30 days postoperatively
Number of readmissions due to urological issues (including urosepsis) | Within the first 30 days postoperatively

OTHER OUTCOMES:
Time from last preoperative micturition to end of surgery. | Patients will be follwed from their last preoperative micturition to end of surgery. Expectably within a mean period of two hours.
Time from last preoperative micturitions to first postoperative bladder catheterization (if relevant). | Patients will be follwed from their last preoperative micturition to their first postoperative bladder catheterization (if relevant). Expectably within a mean period of six to eight hours.
Time from last preoperative micturition to first postoperative, voluntary micturition. | Patients will be follwed from their last preoperative micturition to their first postoperative, voluntary micturition. Expectably within a mean period of fourteen hours.
Time from end of surgery to first postoperative bladder catheterization (if relevant). | Patients will be follwed from end of surgery to their first postoperative bladder catheterization (if relevant). Expectably within a mean period of four to six hours.
Time from end of surgery to first postoperative, voluntary micturition. | Patient will be followed from end of surgery to their first postoperative, voluntary micturition. Expectably within a mean period of twelve hours.

CONTACTS AND LOCATIONS:
Overall Officials: Lars Bjerregaard, MD, Principal Investigator — Rigshospitalet, Copenhagen university, Denmark
Locations (3):
- Denmark (3):
  - Aalborg University Hospital, Farsoe, Farsø
  - Department of Orthopaedics, Gentofte University Hospital, Hellerup
  - Department of Orthopaedics, Vejle Hospital, Vejle